CLINICAL TRIAL: NCT02025881
Title: Phase I / II Study of Sequential High-dose Chemotherapy With Stem Cell Support in Children Younger Than 5 Years of Age With High-risk Medulloblastoma
Brief Title: Study of Sequential High-dose Chemotherapy in Children With High Risk Medulloblastoma
Acronym: HR MB-5
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-004842-14; 2012/1908 (Other: CSET number)
Record Dates: First submitted 2013-12-30; First posted 2014-01-01 (Estimated); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: High-risk Medulloblastoma
MeSH Terms: interventions — EC regimen; Thiotepa; Cyclophosphamide; Busulfan; Irinotecan; Etoposide; Radiotherapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Carboplatin + etoposide then thiotepa then Cyclophosphamide + Busilvex. If insufficient response: TEMIRI + etoposide/radiotherapy + temozolomide
  Interventions: Drug: Carboplatin + etoposide; Drug: Thiotepa; Drug: Cyclophosphamide + Busilvex; Drug: Temozolimide + Irinotecan; Combination Product: Etoposide + radiotherapy; Drug: Temozolomide

INTERVENTIONS:
Drug: Carboplatin + etoposide — Carboplatin 160 mg/m^2 Day 1 to day 5, as an intravenous infusion over 1 hour. Dilution in 5 % glucose saline or sodium chloride 9 mg/ml (0.9%).
  Etoposide 100 mg/m^2 D ay 1 to day 5, as an intravenous infusion over 1 hour. Dilution in physiological saline or 5 % glucose saline while not exceeding a concentration of 0.4 mg/ml etoposide in the infusion bottle.
Drug: Thiotepa — Thiotepa 200 mg/m² Day-3 to day-1, as an intravenously infusion over 1 hour dilution in 200 ml/m^2 of 5% glucose saline or sodium chloride 9 mg/ml (0.9%).
Drug: Cyclophosphamide + Busilvex — Cyclophosphamide:
  * Level 1 20 mg/kg/day
  * Level 2 30 mg/kg/day
  * Level 3 40 mg/kg/day
  * Level 4 50 mg/kg/day
  Busilvex:
  < 9 kgs 0.8 mg/kg/dose -> 3.2 mg/kg/day; 9 à < 16 kgs 0.96 mg/kg/dose -> 3.84 mg/kg/day; 16 à 23 kgs 0.88 mg/kg/dose -> 3.52 mg/kg/day; > 23 à 34 kgs 0.76 mg/kg/dose -> 3.04 mg/kg/day; > 34 kgs -> 0.64 mg/kg/dose.
Drug: Temozolimide + Irinotecan — During 2 cycles of 21 days:
  * Temozolomide: 100 mg/m^2/day PO from Day 1 to Day 5;
  * Irinotecan: 10 mg/m^2/day IV from Day 1 to Day 5 + from Day 8 to Day 12
Combination Product: Etoposide + radiotherapy — * Etoposide: 35 mg/m^2/day PO during 21days
  * Radiotherapy: 1.8 Gy/fraction/day (total dose: 54 Gy)
Drug: Temozolomide — 150 mg/m^2/day PO during 5 days, during 6 cycles of 21 days

SUMMARY:
The trial includes i) the evaluation of the efficacy of a treatment strategy, designed as a phase II trial, and ii) a dose-finding part.

The Phase II trial is an open label, non-randomized, multicentre trial without control group. A Bayesian approach will be used to analyse the EFS, assuming a cure model. We will use three prior distributions of the EFS; (1) an enthusiastic prior distribution, (2) a pessimistic prior distribution, and (3) a non-informative prior distribution. As the patient outcomes in the trial will be recorded, the subsequent distribution of the outcome probability under experimental treatment will be computed by applying Bayes' theorem, which yields an estimated EFS probability with a 95% credibility interval (measure of Bayesian precision). Two interim analyses are planned to monitor the efficacy data (early stopping rules for futility or inefficacy).

The final analysis of efficacy will be made on an intention to treat basis, including all recruited patients, 3 years after recruitment of the last patient.

Due to the uncertainty on the dose of cyclophosphamide that can be given in combination with Busilvex for the last chemotherapy course in patients in complete response after intensification chemotherapy treatment, a dose-finding subtrial will be performed to address this issue (Phase I part). The dose escalation of cyclophosphamide will be performed using the Continual Reassessment Method in a Bayesian framework.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of medulloblastoma with no INI-1 loss
* High risk medulloblastoma defined by at least one of the following conditions:

  * Newly diagnosed classical metastatic medulloblastoma
  * Newly diagnosed anaplastic/large cell medulloblastoma or other unfavourable histology confirmed by review and coordinating investigator
  * Newly diagnosed medulloblastoma with amplification of c-myc or N-myc
* Age at initial biopsy less or equal than 5 years
* Weight compatible with leukapheresis
* Ability to comply with requirements for submission of materials for central review
* Nutritional and general status compatible with this therapy, Lansky play score >/= 30%
* Estimated life expectancy >/=3 months
* No organ toxicity other than neurological symptoms (grade >2 according to NCI-Common Toxicity Criteria v4.0 grading system)
* No prior irradiation or chemotherapy (except Vepesid - CBP)
* Written informed consent from parents or legal guardian
* All patients must be affiliated to a social security regimen or be a beneficiary of the same in order to be included in the study.

Inclusion criteria for the Phase I part of the study:

* Complete response after intensification phase confirmed by central review
* Adequate hepatic and renal function

Exclusion Criteria:

* Desmoplastic medulloblastoma
* Atypical Teratoid rhabdoid tumour
* Uncontrolled active or symptomatic intracranial hypertension
* Patient incapable of undergoing medical follow-up
* Relapse of medulloblastoma

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2013-09-14 (Actual); Primary Completion 2020-10-25 (Actual); Study Completion 2020-10-25 (Actual)

PRIMARY OUTCOMES:
Phase I - Maximum Tolerated Dose | From inclusion to the Dose Limiting Toxicity up to 12 months
  To determine the Maximum Tolerated Dose (MTD) of cyclophosphamide in combination with a fixed dose of Busilvex in children with high-risk medulloblastoma who are in complete response after the intensification phase.
Phase II - Event Free Survival | From inclusion to Event up to 3 years
  To assess the efficacy in terms of Event Free Survival (EFS) of the strategy intended to treat children younger than 5 years of age suffering from high-risk medulloblastoma with sequential high-dose chemotherapy without radiotherapy.

SECONDARY OUTCOMES:
Radiotherapy-free survival without event | From inclusion up to 3 years
Overall Survival | From inclusion up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Dufour, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (13):
- France (13):
  - Gustave Roussy, Villejuif, Val De Marne
  - Institut de Cancérologie de l'Ouest (ICO) - Site Paul Papin, Angers
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - CHU La Timone, Marseille
  - CHU Arnaud de Villeneuve, Montpellier
  - CHU Nancy Brabois, Nancy
  - CHU de Nice - Hôpital L'Archet 2, Nice
  - Institut Curie, Paris
  - Hôpital Américain, Reims
  - CHU Hôpital Sud, Rennes
  - CHRU Hautepierre, Strasbourg
  - Hôpital des enfants, Toulouse